CLINICAL TRIAL: NCT00105846
Title: An Evaluation of Home-Based Telemedicine Services
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEL 20-015
Record Dates: First submitted 2005-03-17; First posted 2005-03-18 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Congestive Heart Failure; Chronic Obstructive Pulmonary Disease; Diabetes
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Home care telemedicine

INTERVENTIONS:
Procedure: Home care telemedicine

SUMMARY:
Tele-home health care, which providers for video interactions between home-based veterans and home care nurses, is a potentially useful adjunct to home care services. However, few randomized trials have been conducted of this technology.

DETAILED DESCRIPTION:
Background:

Tele-home health care, which providers for video interactions between home-based veterans and home care nurses, is a potentially useful adjunct to home care services. However, few randomized trials have been conducted of this technology.

Objectives:

The primary objectives were to determine if tele-home health care patients, compared with patients receiving usual home care, have:1) higher levels of health related quality of life and home care satisfaction; 2) fewer inpatient admissions, hospital stays, and outpatient and emergency room visits; and 3) higher levels of home care access, in terms of the total number of contacts between HBPC nurses and patients.

Methods:

Patients were randomly assigned to the intervention or to the control group. Video tele-health units were installed in patient homes for the intervention group, and control group patients received usual home care services. Baseline and six month follow up surveys included questions on perceived health related quality of life and home care satisfaction. T-tests were used to compare intervention and control group members in terms of six month changes in health related quality of life and satisfaction with home care. Multivariate analyses were used to assess group differences in six month health care service use, with prior service use and survival included as covariates.

Status:

The study is completed, with a final enrollment of 37 patients. Three study manuscrip[ts have been completed (two published and one under review).

ELIGIBILITY:
Inclusion Criteria:

Patients must be enrolled in the home care program at the Indianapolis VAMC and have at least: (a) 6 outpatient visits, one hospitalization, or 2 or more emergency room visits in the last twelve months, (b) a care plan specifying two or more skilled nursing visits per month, (c) an expected need for future home care visits for at least one month.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith P. Hopp, PhD MA MSW, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Nebraska

REFERENCES:
- [Result] Hopp F, Woodbridge P, Subramanian U, Copeland L, Smith D, Lowery J. Outcomes associated with a home care telehealth intervention. Telemed J E Health. 2006 Jun;12(3):297-307. doi: 10.1089/tmj.2006.12.297. PMID 16796497
- [Result] Subramanian U, Hopp F, Lowery J, Woodbridge P, Smith D. Research in home-care telemedicine: challenges in patient recruitment. Telemed J E Health. 2004 Summer;10(2):155-61. doi: 10.1089/tmj.2004.10.155. PMID 15319045
- [Result] Hopp F, Woodbridge P, Subramanian U, Copeland L, Smith D. Home telehealth's role in diabetes case management. Telemedicine journal and e-health : the official journal of the American Telemedicine Association. 2005 Apr 1; 11:220.